CLINICAL TRIAL: NCT03963622
Title: Careful Ventilation in Acute Respiratory Distress Syndrome
Brief Title: Careful Ventilation in Acute Respiratory Distress Syndrome (COVID-19 and Non-COVID-19)
Acronym: CAVIARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other); Applied Health Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1765
Record Dates: First submitted 2019-05-06; First posted 2019-05-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: ARDS
Keywords: Ventilation; ARDS; Airway closure; Lung recruitment; COVID-19; Basket trial
MeSH Terms: conditions — Respiratory Aspiration; COVID-19 | interventions — Respiratory Mechanics

STUDY DESIGN:
Intervention Model Description: This study is also a basket design, which examines a single intervention in multiple disease populations. This basket trial consists of an identical 2-arm mechanical ventilation protocol implemented in two different study populations (patients with COVID-19-induced ARDS, and patients with all ARDS not induced by COVID-19). The protocol and procedures are identical between the two study populations in this basket trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard ventilation strategy.
  Interventions: Other: Standard Ventilation Strategy
- Respiratory Mechanics (Experimental): The goal of this arm is to individualize tidal volume (VT) and PEEP according to respiratory mechanics.
  Interventions: Other: Respiratory Mechanics

INTERVENTIONS:
Other: Respiratory Mechanics — Different maneuvers based on respiratory mechanics will be assessed at the bedside and will be used to individualize ventilator parameters. Recruitability will be assessed with a one breath decremental PEEP maneuver, and search for airway closure with a low-flow pressure volume or pressure-time curve. If the patient has airway closure, the minimal PEEP will be set at the airway opening pressure to avoid closure. If the patient is considered recruitable, the goal is to set PEEP at or above 15cmH20 to maximize alveolar recruitment, until the plateau pressure reaches the safety limit. Volume control ventilation at 6ml·kg-1 will be used.
  Once spontaneous breathing has started, the occlusion pressure (P0.1) will be maintained within targets.
  Arms: Respiratory Mechanics
Other: Standard Ventilation Strategy — Patients randomized to the control arm will receive standard care. The PEEP is adjusted for oxygenation based on a PEEP-FiO2 table, either the low PEEP-FiO2 or the high PEEP-FiO2 table. Volume targeted ventilation with initial VT 6 mL·kg-1 and Plateau pressure at 30 cmH2O or below, targeting PaO2 60-80 or SpO2 90-95%, adjusted as per the protocol. Pressure-support ventilation is at physician's discretion, but recommended when FiO2 <60%, and is titrated VT 6-8 mL·kg-1.
  Arms: Control

SUMMARY:
This is a multicenter randomized controlled clinical trial with an adaptive design assessing the efficacy of setting the ventilator based on measurements of respiratory mechanics (recruitability and effort) to reduce Day 60 mortality in patients with acute respiratory distress syndrome (ARDS).

The CAVIARDS study is also a basket trial; a basket trial design examines a single intervention in multiple disease populations. CAVIARDS consists of an identical 2-arm mechanical ventilation protocol implemented in two different study populations (COVID-19 and non-COVID-19 patients). As per a typical basket trial design, the operational structure of both the COVID-19 substudy (CAVIARDS-19) and non-COVID-19 substudy (CAVIARDS-all) is shared (recruitment, procedures, data collection, analysis, management, etc.).

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is a major public health problem affecting approximately 10% of patients in the intensive care unit (ICU) and 23% of all patients on a breathing machine (mechanical ventilator). The short-term mortality of patients with ARDS is approximately 40% and better ventilation of these patients has the greatest potential to improve outcomes.

The lungs in patients with ARDS are severely inflamed which reduces lung volume and their ability to stretch, making ventilation difficult and dangerous. However, mechanical ventilation is the mainstay of supportive therapy. Although it is life-saving, it can also can generate secondary injury and inflammation, called ventilator-induced lung injury (VILI). The investigators know that inadequate mechanical ventilation worsens outcomes but are uncertain of the optimal way to manage ventilators at the bedside.

Furthermore, ARDS is challenging because there is no treatment for the alveolar-capillary leak characterizing this syndrome; aside from treating the underlying cause, the only supportive therapy is mechanical ventilation. This is specially the case for COVID-19 induced ARDS. Despite best practices, over-distension of the lung or inappropriate positive end expiratory pressure (PEEP) is common. Finally, once spontaneous breathing has resumed and is assisted by the ventilator, an additional phenomenon occurs, called patient self-inflicted lung injury. The drive for breathing in many patients is stimulated by lung inflammation, and strong breathing efforts can generate high distending pressures, causing lung (and systemic) inflammation and organ damage. Whether the management of COVID-19 induced ARDS should differ from all other ARDS has been debated at length but has no clear response

Recent advances in our understanding of bedside physiology (airway closure, recruitability, lung distension, respiratory drive) can now be applied for an individual titration of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 y
2. Moderate or severe ARDS (PaO2/FiO2 ≤ 200 mmHg) within 48 h of meeting Berlin ARDS criteria (Patients who were eligible at the time of screening and whose PaO2/FiO2 became > 200 mm Hg under prone positioning when starting the protocol remained eligible)

Exclusion Criteria:

1. Received continuous mechanical ventilation > 7 days
2. Known or clinically suspected elevated intracranial pressure (>18mmHg) necessitating strict control of PaCO2
3. Known pregnancy
4. Broncho-pleural fistula
5. Severe liver disease (Child-Pugh Score ≥ 10)
6. BMI >40kg/m2
7. Anticipating withdrawal of life support and/or shift to palliation as the goal of care
8. Patient is receiving ECMO at time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
All-cause 60-day mortality | 60 days
  The lack of an appropriate surrogate endpoint, and the high baseline mortality rate mandate a multicentre RCT to determine the mortality effects of setting the ventilator based on recruitability and effort compared with conventional ventilation.

SECONDARY OUTCOMES:
Duration of ventilation | May exceed 60 days
  Duration of ventilation in days
Duration of ICU and hospital stay | May exceed 60 days
  Duration of ICU and hospital stay in days
Number of patients with organ dysfunction | Day 1-7, 14, 21, 28
  Organ dysfunction as per the SOFA score
Number of patients with barotrauma | Up to 60 days
  Barotrauma defined as new onset of pneumothorax
Mortality at ICU discharge, 28 days, and hospital discharge | Up to date of ICU discharge, 28 days, and hospital discharge
  Mortality

OTHER OUTCOMES:
The change in biomarker expression | Baseline, 24 and 72 hours
  Biomarkers include interleukin 6 (IL-6), interleukin 8 (IL-8), tumor necrosis factor receptor 1 (TNFr1), soluble receptor of the advanced glycation end products (sRAGE), and surfactant protein D (SPD). All measured in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, MD, Principal Investigator — Unity Health Toronto
Locations (33):
- New York University Grossman School of Medicine, New York, New York, United States
- Argentina (6):
  - Centro de Educación Médica e Investigaciones Clínicas Dr Norberto Quirno (CEMIC), Buenos Aires
  - Complejo Médico Policía Federal Argentina Churruca Visca, Buenos Aires
  - Hospital Británico de Buenos Aires, Buenos Aires
  - Sanatorio Anchorena Recoleta, Buenos Aires
  - Sanatorio Mater Dei, Buenos Aires
  - Sanatorio Anchorena San Martín, San Martín
- Canada (3):
  - St. Michael's Hospital, Toronto
  - Toronto General Hospital, Toronto
  - Toronto Western Hospital, Toronto
- Pontificia Universidad Católica de Chile, Santiago, Chile
- France (16):
  - CHU Amiens-Picardie, Amiens
  - Centre hospitalier universitaire d'Angers, Angers
  - CH Victor Dupouy, Argenteuil
  - CH de Beauvais, Beauvais
  - CHU Bordeaux - Haut Leveque, Bordeaux
  - Hopital de la Cavale Blanche - CHRU Brest, Brest
  - CH de Cholet, Cholet
  - Hopital Intercommunal de Creteil, Créteil
  - CHU Grenoble-Alpes, Grenoble
  - Hopital Roger Salengro - CHU Lille, Lille
  - Groupe Hospitalier de la Region de Mulhouse et Sud Alsace, Mulhouse
  - Hopital de l'Archet 1 - CHU de Nice, Nice
  - Hopital Europeen Georges-Pompidou, Paris
  - CHU de Poitiers - La Miletrie, Poitiers
  - CH Bretagne Atlantique Vannes-Auray, Vannes
  - HIA Robert Picque, Villenave-d'Ornon
- Italy (3):
  - Arcispedale Sant'Anna, Ferrara
  - University of Foggia, Foggia
  - Policlinico Universitario Agostino Gemelli IRCCS, Rome
- OLVG, Amsterdam, North Holland, Netherlands
- Spain (2):
  - L'Hospital de la Santa Creu i Sant Pau, Barcelona
  - Vall d'Hebron University Hospital, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
The final anonymized trial dataset will be available on reasonable written request to the principal investigator one year after publication of the main manuscript.

REFERENCES:
- [Derived] Villalba DS, Matesa A, Boni S, Gutierrez FJ, Moracci R, Plotnikow GA. Impact of High-Flow Nasal Cannula Oxygen Therapy on the Pressure of the Airway System in Humans. Respir Care. 2025 Jan;70(1):10-16. doi: 10.1089/respcare.12082. PMID 39964860
- See also: Study website — https://studykeepr.com/caviards